CLINICAL TRIAL: NCT01390909
Title: Clinical and Economic Burden of Uncontrolled Epilepsy: Analyses From a Medicaid Database and a Private Health Plan Database
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113917
Record Dates: First submitted 2011-07-07; First posted 2011-07-11 (Estimated); Results first posted 2012-02-14 (Estimated); Last update posted 2012-10-08 (Estimated); Status verified 2012-06

CONDITIONS: Epilepsy
Keywords: epilepsy; anti-epileptic drug; polytherapy; adherence; Medicaid
MeSH Terms: conditions — Epilepsy | interventions — Anticonvulsants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Medicaid patients with uncontrolled epilepsy: Database records for patients with 2 or more consecutive changes in anti-epileptic drug (AED) therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or emergency department (ED) visits within the 365 days
  Interventions: Drug: Anti-epileptic drug (AED)
- Medicaid patients with well-controlled epilepsy: Database records for patients with an epilepsy diagnosis but no AED change and no epilepsy-related inpatient or ED visits
  Interventions: Drug: Anti-epileptic drug (AED)
- Medicaid patients with intermediate epilepsy: Database records for patients who are not classified as uncontrolled or well-controlled
  Interventions: Drug: Anti-epileptic drug (AED)
- Patients in a private health plan with uncontrolled epilepsy: Database records for patients with 2 or more consecutive changes in AED therapy occuring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or ED visits within 365 days
  Interventions: Drug: Anti-epileptic drug (AED)
- Patients in a private health plan with well-controlled epileps: Database records for patients with an epilepsy diagnosis but no AED change and no epilepsy-related inpatient or ED visits
  Interventions: Drug: Anti-epileptic drug (AED)
- Patients in a private health plan with intermediate epilepsy: Database records for patients who are not classified as uncontrolled or well-controlled
  Interventions: Drug: Anti-epileptic drug (AED)

INTERVENTIONS:
Drug: Anti-epileptic drug (AED) — Prescription claim for at least one AED including lamotrigine, tiagabine, pregabalin, ethosuximide, lacosamide, phenytoin, carbamazepine, valproic acid, felbamate, levetiracetam, zonisamide, primidone, oxcarbazepine, vigabatrin, phenobarbital, gabapentin, topiramate.
  Other Names: Mysoline® is a registered trademark of Valeant Pharmaceuticals; Neurotin® is registered trademark of Pfizer; Inc; Vimpat® is a registered trademark of UCB Pharma; Tegretol® is a registered trademark of Novartis Pharmaceuticals; Trileptal® is a registered trademark of Novartis Pharmaceuticals; Sabril® is a registered trademark of Lundbeck Inc; Felbatol® is a registered trademark of MedPointe; Topamax® is a registered trademark of Ortho-McNeill-Janssen Pharmaceuticals; Depakote® is a registered trademark of Abbott Laboratories; Zonegran® is a registered trademark of Dainippon Pharmaceutical C. Ltd.; Gabatril® is a registered trademark of Cephalon; Keppra® is registered trademark of UCB Pharma; Zarontin® is a registered trademark of Pfizer; Lamictal® is a registered trademark of GlaxoSmithKline; Luminal® is a registered trademark of Abbott Laboratories; Dilantin® is a registered trademark of Pfizer; Lyrica is registered trademark of Pfizer

SUMMARY:
Antiepileptic drugs (AEDs) are the main therapeutic option for patients with epilepsy; however, complete seizure control remains elusive for many patients. Uncontrolled or refractory epilepsy is associated with a higher risk of mortality, physical injuries, and depression or anxiety compared with patients with controlled epilepsy. Higher resource utilization for patients with poor control is likely to be associated with higher economic costs. While diagnostic criteria for uncontrolled epilepsy are debated by neurologists, recent studies suggest that a diagnosis of uncontrolled epilepsy requires 1.) at least one seizure per month and 2.) a history of drug failures.

The objective of this study is to identify patients with uncontrolled epilepsy in both a Medicaid database and a private health plan database, to describe patient characteristics and AED treatment patterns between cohorts of patients with uncontrolled versus well-controlled epilepsy, and to evaluate the economic burden of uncontrolled versus well-controlled epilepsy.

For this evaluation, the data sources are medical and pharmacy claims in Medicaid databases from Florida (Third quarter 1997 to second quarter 2008), Iowa (First quarter 1998 to second quarter 2006), Kansas (First quarter 2001 to second quarter 2009), Missouri (First quarter 1997 to second quarter 2008) and New Jersey (First quarter 1997 to fourth quarter 2008) and medical and pharmacy claims in an private health plan database.

The study design is a retrospective, longitudinal, matched-cohort study. Eligible patient records will be assigned to one of three mutually-exclusive cohorts: uncontrolled epilepsy (at least 2 consecutive changes in AED therapy in at least 30 days, and at least 1 epilepsy-related inpatient or emergency department (ED) visit within 365 days), well-controlled epilepsy (no AED changes and no epilepsy-related inpatient or ED visits), and intermediate epilepsy (not classified as uncontrolled or well-controlled).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the initiation of anti-epileptic drug (AED) treatment as noted in the database
* A record of at least one medical visit with a diagnosis of epilepsy (ICD-9-CM 345.xx) or at least two diagnoses of non-febrile convulsions (ICD-9-CM 780.30 or 780.39) occuring more than 30 days apart
* At least one pharmacy claim for an anti-epileptic drug (AED)
* Continuous enrollment throughout the observation period (minimum of 365 days). Patients with gaps in Medicaid enrollment will be observed only during their period of continuous enrollment, provided that all the above criteria are met

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The electronic records from adult patients with epilepsy who are enrolled in Medicaid in Florida, Iowa, Kansas, Missouri or New Jersey or in a private health plan database. Patient records will be classified into one of three mutually-exclusive cohorts: uncontrolled epilepsy, well-controlled epilepsy, and intermediate epilepsy (not classified as uncontrolled or well-controlled).
Sampling Method: Non-Probability Sample
Enrollment: 12386 (Actual)
Dates: Start 2010-05; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Groups:
- Medicaid, Well Controlled: Database records for participants with an epilepsy diagnosis but no AED change and no epilepsy-related inpatient or ED visits
- Medicaid, Uncontrolled: Database records for participants with 2 or more consecutive changes in AED therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or ED visits within the next 365 days. This arm represents all participant records that met the criteria for uncontrolled epilepsy. Participants in the Medicaid, Uncontrolled, Subgroup were matched with participant records in the Medicaid, well-controlled cohort.
- Medicaid, Intermediate; Private, Intermediate: Database records for participants who are not classified as uncontrolled or well controlled
- Private, Well Controlled: Database records for participants with an epilepsy diagnosis but no AED change and no epilepsy-related inpatient or ED visit
- Private, Uncontrolled: Database records for participants with 2 or more consecutive changes in AED therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or ED visit within the next 365 days. This arm represents all participant records that met the criteria for uncontrolled epilepsy. Participants in the Medicaid, Uncontrolled, Subgroup were matched with participant records in the Medicaid, well-controlled cohort.
Period: Overall Study
Arm/Group | Medicaid, Well Controlled | Medicaid, Uncontrolled | Medicaid, Intermediate | Private, Well Controlled | Private, Uncontrolled | Private, Intermediate
Started | 3454 | 3552 | 3552 | 602 | 613 | 613
Participants in Subgroup | 0 | 3454 | 0 | 0 | 602 | 0
Completed | 3454 | 3552 | 3552 | 602 | 613 | 613
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Medicaid, Uncontrolled: Database records for participants with 2 or more consecutive changes in AED therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or ED visits within the next 365 days. This arm represents all participant records that met the criteria for uncontrolled epilepsy. Participants in the Medicaid, Uncontrolled, Subgroup (3454 participants) were matched with participant records in the Medicaid, well-controlled cohort.
- Private, Well Controlled: Database records for participants with an epilepsy diagnosis but no AED change and no epilepsy-related inpatient or ED visits
- Private, Uncontrolled: Database records for participants with 2 or more consecutive changes in AED therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or ED visits within the next 365 days. This arm represents all participant records that met the criteria for uncontrolled epilepsy. Participants in the Medicaid, Uncontrolled, Subgroup (602 participants) were matched with participant records in the Medicaid, well-controlled cohort.
- Total: Total of all reporting groups
Arm/Group | Medicaid, Well Controlled | Medicaid, Uncontrolled | Medicaid, Intermediate | Private, Well Controlled | Private, Uncontrolled | Private, Intermediate | Total
Number analyzed (Participants) | 3454 | 3552 | 3552 | 602 | 613 | 613 | 12386
Age Continuous [Mean (Standard Deviation); unit: Years] — For the total population and the subgroup total population, a weighted average of the individual study group means and number of participants was used. The standard deviation (SD) is the SD of the study group means.
  Years
    Overall Study | 41.5 (15.4) | 41.3 (14.1) | 41.2 (14.6) | 54.2 (17.1) | 54.1 (17.3) | 54.6 (16.7) | 43.2 (6.5)
    Subgroup | NA (NA) — There are no subgroup participants. | 41.4 (14.2) | NA (NA) — There are no subgroup participants. | NA (NA) — There are no subgroup participants. | 54.0 (17.4) | NA (NA) — There are no subgroup participants. | 43.3 (6.3)
Sex/Gender, Customized [Number; unit: Participants]
  Female, Overall Study | 2106 | 2171 | 2159 | 341 | 351 | 332 | 7460
  Male, Overall Study | 1348 | 1381 | 1393 | 261 | 262 | 281 | 4926
  Female, Subgroup | NA — There are no subgroup participants. | 2091 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 345 | NA — There are no subgroup participants. | 2436
  Male, Subgroup | NA — There are no subgroup participants. | 345 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 257 | NA — There are no subgroup participants. | 602
Number of Days of Observation [Mean (Standard Deviation); unit: days of observation] — For the total population and subgroups, a weighted average of the individual study group means and number of participants was used. The SDs reflect the SDs of the study group means.
  days of observation
    Overall Study | 2184 (1181) | 2296 (1132) | 2502 (1124) | 1572 (847) | 1478 (749) | 1739 (792) | 2221 (385)
    Subgroup | NA (NA) — There are no subgroup participants. | 2290 (1133) | NA (NA) — There are no subgroup participants. | NA (NA) — There are no subgroup participants. | 1485 (751) | NA (NA) — There are no subgroup participants. | 2170.5 (402.5)
Charlson Comorbidity Index (CCI) Scores [Mean (Standard Deviation); unit: scores on a scale] — The Charlson Comorbidity Index estimates 10-year mortality risk. Scores range from 0 - 37, with a lower score indicating a higher chance of survival. For the total population and the subgroup, a weighted average of the study group means was used. The standard deviation (SD) is the SD of the study group means.
  scores on a scale
    Overall Study | 0.98 (1.83) | 1.09 (1.84) | 1.00 (1.78) | 1.13 (1.65) | 1.32 (1.91) | 1.20 (1.82) | 1.05 (0.11)
    Subgroup | NA (NA) — There are no subgroup participants. | 1.08 (1.83) | NA (NA) — There are no subgroup participants. | NA (NA) — There are no subgroup participants. | 1.29 (1.88) | NA (NA) — There are no subgroup participants. | 1.11 (1.66)
Number of participant records with diagnosis codes for the indicated diseases or disorders [Number; unit: participant records]
  Alzheimer's Disease, Overall Study | 94 | 93 | 84 | 12 | 20 | 19 | 322
  Alzheimer's Disease Subgroup | NA — There are no subgroup participants. | 93 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 20 | NA — There are no subgroup participants. | 113
  Brain Tumor, Overall Study | 53 | 63 | 40 | 38 | 50 | 43 | 287
  Brain Tumor, Subgroup | NA — There are no subgroup participants. | 62 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 44 | NA — There are no subgroup participants. | 106
  Meningitis, Overall Study | 12 | 16 | 13 | 11 | 10 | 6 | 68
  Meningitis, Subgroup | NA — There are no subgroup participants. | 15 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 9 | NA — There are no subgroup participants. | 24
  Migraine, Overall Study | 198 | 262 | 262 | 41 | 42 | 35 | 840
  Migraine, Subgroup | NA — There are no subgroup participants. | 239 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 41 | NA — There are no subgroup participants. | 280
  Stroke, Overall Study | 267 | 303 | 264 | 123 | 134 | 154 | 1245
  Stroke, Subgroup | NA — There are no subgroup participants. | 302 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 128 | NA — There are no subgroup participants. | 430
  Anxiety Disorders, Overall Study | 356 | 447 | 440 | 32 | 41 | 28 | 1344
  Anxiety Disorders, Subgroup | NA — There are no subgroup participants. | 410 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 38 | NA — There are no subgroup participants. | 448
  Bipolar Disorder, Overall Study | 428 | 439 | 472 | 22 | 18 | 15 | 1394
  Bipolar Disorder, Subgroup | NA — There are no subgroup participants. | 397 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 17 | NA — There are no subgroup participants. | 414
  Depression, Overall Study | 821 | 890 | 897 | 90 | 95 | 102 | 2895
  Depression, Subgroup | NA — There are no subgroup participants. | 833 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 90 | NA — There are no subgroup participants. | 923
  Psychosis, Overall Study | 809 | 794 | 816 | 62 | 65 | 65 | 2611
  Psychosis, Subgroup | NA — There are no subgroup participants. | 754 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 65 | NA — There are no subgroup participants. | 819
  Personality Disorder, Overall Study | 951 | 1062 | 1024 | 51 | 68 | 58 | 3214
  Personality Disorder, Subgroup | NA — There are no subgroup participants. | 1001 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 67 | NA — There are no subgroup participants. | 1068
  Mental Retardation, Overall Study | 482 | 322 | 434 | 5 | 11 | 8 | 1262
  Mental Retardation, Subgroup | NA — There are no subgroup participants. | 312 | NA — There are no subgroup participants. | NA — There are no subgroup participants. | 11 | NA — There are no subgroup participants. | 323

OUTCOME MEASURES:

1. Primary Outcome: Average Annualized Costs
Description: Average annualized overall healthcare costs and epilepsy-related healthcare costs were calculated for each treatment group. Epilepsy-related costs were those with a code for epilepsy. ED, Emergency Department; AMC, All Medical Costs; Ep Rel, Epilepsy Related. United States dollars were consumer price index adjusted for 2009.
Time Frame: 1 year
Population: For Arms 1 - 4, Medicaid-enrolled participants with uncontrolled epilepsy (see Arm Descriptions for Arm Title 1 and Arm Title 3) or matched participants with well-controlled or intermediate epilepsy. For Arms 5 - 8, privately-insured participants with uncontrolled epilepsy or matched participants with well-controlled or intermediate epilepsy.
Measure: Mean (Standard Deviation); unit: United States dollars
Groups:
- Medicaid, Uncontrolled, Subgroup: Database records for participants with 2 or more consecutive changes in anti-epileptic drug (AED) therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or emergency department (ED) visits within the next 365 days. This subgroup was matched with participant records in the Medicaid, well-controlled cohort
- Medicaid, Uncontrolled: Database records for participants with 2 or more consecutive changes in AED therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or ED visits within the next 365 days. This arm represents all participant records that met the criteria for uncontrolled epilepsy
- Private, Uncontrolled, Subgroup: Database records for participants with 2 or more consecutive changes in AED therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or ED visit within the next 365 days. This subgroup was matched with participant records in the private, well-controlled cohort.
- Private, Uncontrolled: Database records for participants with 2 or more consecutive changes in AED therapy occurring at least 30 days apart and followed by 1 or more epilepsy-related inpatient or ED visit within the next 365 days. This arm represents all participant records that met the criteria for uncontrolled epilepsy.
Arm/Group | Medicaid, Uncontrolled, Subgroup | Medicaid, Well Controlled | Medicaid, Uncontrolled | Medicaid, Intermediate | Private, Uncontrolled, Subgroup | Private, Well Controlled | Private, Uncontrolled | Private, Intermediate
Number analyzed (Participants) | 3454 | 3454 | 3552 | 3552 | 602 | 602 | 613 | 613
United States dollars
  AEDs | 1352 (4580) | 462 (2072) | 1357 (4590) | 1050 (4297) | 1697 (3979) | 639 (2248) | 1713 (3989) | 1299 (3949)
  Non-AEDs | 5615 (15730) | 3657 (11702) | 5725 (16016) | 4801 (15357) | 4497 (11374) | 3096 (10692) | 4587 (11972) | 3883 (9436)
  Hospitalizations; AMC | 6902 (31181) | 958 (9518) | 7041 (31499) | 3513 (22265) | 11308 (62399) | 1697 (12292) | 12357 (84898) | 5858 (37310)
  ED Visits; AMC | 400 (1496) | 97 (731) | 421 (1661) | 242 (1371) | 586 (4392) | 76 (804) | 603 (4422) | 254 (2898)
  Outpatient Visits; AMC | 2416 (11759) | 1258 (9953) | 2466 (11829) | 1804 (11649) | 5757 (24888) | 3061 (13353) | 5771 (24883) | 5780 (37154)
  Neurology Visits; AMC | 86 (850) | 21 (425) | 86 (839) | 52 (666) | 556 (4306) | 175 (1593) | 566 (4352) | 442 (4263)
  Other Healthcare Services; AMC | 22022 (106033) | 23202 (103595) | 22113 (107291) | 23428 (119218) | 1008 (5428) | 436 (4444) | 1026 (5472) | 645 (3910)
  Hospitalizations; Ep Rel | 4102 (19775) | NA (NA) — None of the participants in this study arm incurred the indicated type of healthcare encounter during the study period. | 4135 (19915) | 1702 (13344) | 6700 (48095) | NA (NA) — None of the participants in this study arm incurred the indicated type of healthcare encounter during the study period. | 7646 (70525) | 2413 (23487)
  ED Visits; Ep Rel | 109 (610) | NA (NA) — None of the participants in this study arm incurred the indicated type of healthcare encounter during the study period. | 111 (616) | 46 (540) | 152 (972) | NA (NA) — None of the participants in this study arm incurred the indicated type of healthcare encounter during the study period. | 153 (968) | 39 (635)
  Outpatient Visits; Ep Rel | 467 (2218) | 68 (490) | 469 (2239) | 248 (1660) | 703 (3072) | 179 (1042) | 702 (3082) | 479 (6624)
  Neurology Visits; Ep Rel | 60 (712) | 9 (143) | 59 (703) | 33 (472) | 235 (1797) | 68 (577) | 237 (1845) | 165 (1670)
  Other Healthcare Costs; Ep Rel | 1502 (14424) | 754 (10724) | 1475 (14265) | 1273 (14072) | 103 (752) | 17 (204) | 102 (746) | 42 (472)
  Total Healthcare Costs; AMC | 38708 (114904) | 29635 (105644) | 39123 (116204) | 34839 (123866) | 24853 (81299) | 9005 (28038) | 26057 (100777) | 17719 (69241)
Statistical Analysis 1: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Prescription Drug Costs, AEDs; Ordinary least squares regression was used to adjust differences. Covariates were gender, age, region, comorbidities, baseline treatment, and costs; Median Difference (Final Values) = 849, 95% CI 2-sided [786 to 921] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 2: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Prescription Drug Costs, nonAEDs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 1879, 95% CI 2-sided [1636 to 2112] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 3: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Hospitalizations, All Medical Costs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 5681, 95% CI 2-sided [5257 to 6077] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 4: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Emergency Department Visits, All Medical Costs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 273, 95% CI 2-sided [251 to 295] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 5: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Outpatient Services, All Medical Costs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 1021, 95% CI 2-sided [819 to 1211] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 6: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Neurologist Visits, All Medical Costs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 60, 95% CI 2-sided [48 to 72] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 7: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p = 0.0080, Ordinary Least Squares Regression — Adjusted Cost Differences in Other Healthcare Services, All Medical Costs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 2555, 95% CI 2-sided [834 to 4281] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 8: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Hospitalizations; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4041, 95% CI 2-sided [3776 to 4305] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 9: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Emergency Department Visits; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 105, 95% CI 2-sided [97 to 114] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 10: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Outpatient Services; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 384, 95% CI 2-sided [358 to 413] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 11: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Neurologist Visits; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 47, 95% CI 2-sided [40 to 56] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 12: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Other Epilepsy-Related Healthcare Costs; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 892, 95% CI 2-sided [584 to 1192] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 13: Comparison: Medicaid, Uncontrolled, Subgroup vs Medicaid, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Total Healthcare Costs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 12258, 95% CI 2-sided [10482 to 14083] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 14: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Prescription Drug Costs, AEDs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 322, 95% CI 2-sided [245 to 398]
Statistical Analysis 15: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Prescription Drug Costs, non-AEDs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 841, 95% CI 2-sided [556 to 1078]
Statistical Analysis 16: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Hospitalizations, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 3248, 95% CI 2-sided [2790 to 3714]
Statistical Analysis 17: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Emergency Department Visits, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 164, 95% CI 2-sided [138 to 190]
Statistical Analysis 18: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Outpatient Services, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Median Difference (Final Values) = 628, 95% CI 2-sided [409 to 819]
Statistical Analysis 19: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Neurologist Visits, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 29, 95% CI 2-sided [18 to 42]
Statistical Analysis 20: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p = 0.7628, Ordinary Least Squares Regression — Adjusted Cost Differences in Other Healthcare Services, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 235, 95% CI 2-sided [-1367 to 1798]
Statistical Analysis 21: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Hospitalizations; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2306, 95% CI 2-sided [2016 to 2603] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 22: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Emergency Department Visits; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 63, 95% CI 2-sided [52 to 74] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 23: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Outpatient Services; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 211, 95% CI 2-sided [179 to 245] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 24: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Neurologist Visits; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 23, 95% CI 2-sided [15 to 33] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 25: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p = 0.0581, Ordinary Least Squares Regression — Adjusted Cost Differences in Other Epilepsy-Related Healthcare Costs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 277, 95% CI 2-sided [-19 to 581] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 26: Comparison: Medicaid, Uncontrolled vs Medicaid, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Total Healthcare Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 5437, 95% CI 2-sided [3672 to 7142]
Statistical Analysis 27: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Prescription Drug Costs, AEDs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 1019, 95% CI 2-sided [836 to 1191]
Statistical Analysis 28: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Prescription Drug Costs, Non-AEDs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Median Difference (Final Values) = 1047, 95% CI 2-sided [564 to 1486]
Statistical Analysis 29: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Hospitalizations; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Median Difference (Final Values) = 9128, 95% CI 2-sided [7346 to 11125]
Statistical Analysis 30: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Emergency Department Visits; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 459, 95% CI 2-sided [326 to 622]
Statistical Analysis 31: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Outpatient Services; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Median Difference (Final Values) = 2427, 95% CI 2-sided [1587 to 3290]
Statistical Analysis 32: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Neurologists Visits; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Median Difference (Final Values) = 357, 95% CI 2-sided [225 to 525]
Statistical Analysis 33: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Other Healthcare Services; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Median Difference (Final Values) = 502, 95% CI 2-sided [234 to 768]
Statistical Analysis 34: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Hospitalizations; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 6483, 95% CI 2-sided [5329 to 7927] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 35: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Emergency Department Visits; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 150, 95% CI 2-sided [112 to 199] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 36: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Outpatient Services; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 516, 95% CI 2-sided [401 to 645] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 37: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Epilepsy-Related Neurologist Visits; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 158, 95% CI 2-sided [97 to 231] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 38: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Other Epilepsy-Related Healthcare Costs; [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = 83, 95% CI 2-sided [58 to 113] — Confidence intervals were calculated using a nonparametric bootstrap with 999 replications
Statistical Analysis 39: Comparison: Private, Uncontrolled, Subgroup vs Private, Well Controlled; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Total Healthcare Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 14582, 95% CI 2-sided [12019 to 17097]
Statistical Analysis 40: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Prescription Drug Costs, AEDs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 420, 95% CI 2-sided [210 to 630]
Statistical Analysis 41: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Prescription Drug Costs, Non-AEDs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 658, 95% CI 2-sided [217 to 1131]
Statistical Analysis 42: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Hospitalizations, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 6040, 95% CI 2-sided [3442 to 8795]
Statistical Analysis 43: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p = 0.0020, Ordinary Least Squares Regression — Adjusted Cost Differences in Emergency Department Visits, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 268, 95% CI 2-sided [81 to 425]
Statistical Analysis 44: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p = 0.9670, Ordinary Least Squares Regression — Adjusted Cost Differences in Outpatient Services, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = -40, 95% CI 2-sided [-991 to 944]
Statistical Analysis 45: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p = 0.2563, Ordinary Least Squares Regression — Adjusted Cost Differences in Neurologist Visits, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 97, 95% CI 2-sided [-77 to 302]
Statistical Analysis 46: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p = 0.0100, Ordinary Least Squares Regression — Adjusted Cost Differences in Other Healthcare Services, All Medical Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 328, 95% CI 2-sided [90 to 588]
Statistical Analysis 47: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Hospitalizations, Epilepsy-Related; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 4984, 95% CI 2-sided [3168 to 7335]
Statistical Analysis 48: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Emergency Department Visits, Epilepsy-Related; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 112, 95% CI 2-sided [70 to 166]
Statistical Analysis 49: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p = 0.01, Ordinary Least Squares Regression — Adjusted Cost Differences in Outpatient Services, Epilepsy-Related; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 236, 95% CI 2-sided [70 to 403]
Statistical Analysis 50: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p = 0.1061, Ordinary Least Squares Regression — Adjusted Cost Differences in Neurologist Visits, Epilepsy-Related; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 65, 95% CI 2-sided [-22 to 145]
Statistical Analysis 51: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Other Healthcare Services, Epilepsy-Related; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 58, 95% CI 2-sided [28 to 93]
Statistical Analysis 52: Comparison: Private, Uncontrolled vs Private, Intermediate; Test type: Superiority or Other; p < 0.0001, Ordinary Least Squares Regression — Adjusted Cost Differences in Total Healthcare Costs; Covariates were gender, age, region, comorbidities, AEDs and non-AEDs known to increase seizure risk and baseline costs; Mean Difference (Final Values) = 7673, 95% CI 2-sided [4571 to 10989]

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | Medicaid, Uncontrolled, Subgroup | Medicaid, Well Controlled | Medicaid, Uncontrolled | Medicaid, Intermediate | Private, Uncontrolled, Subgroup | Private, Well Controlled | Private, Uncontrolled | Private, Intermediate
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.